CLINICAL TRIAL: NCT03525210
Title: An Open-label Phase III Study to Investigate the Safety, Tolerability and Immunogenicity of a Nine-valent Human Papillomavirus (HPV) Vaccine (Gardasil®9) in Solid Organ Transplant Recipients and HIV-infected Patients
Brief Title: Study of Safety, Tolerability and Immunogenicity of Gardasil®9 in Immunocompromised Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 503-IC; NCT03482739 (obsolete NCT alias)
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Human Papilloma Virus; Hiv; Organ Transplants
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIV patients (Other): All HIV patients will receive the study vaccines
  Interventions: Biological: 9-valent HPV vaccine
- SOT patients (Other): All SOT patients will receive the study vaccines
  Interventions: Biological: 9-valent HPV vaccine

INTERVENTIONS:
Biological: 9-valent HPV vaccine — Vaccination
  Other Names: Gardasil9

SUMMARY:
Patients with immunodeficiencies are at increased risk of developing persistent HPV infection and as such HPV-related disease (genital warts and cancer).

In this study HIV-patients and SOT-patients will receive 3 doses of Gardasil®9. Safety, tolerability and immunogenicity will be evaluated up to one month following the 3rd and last dose of Gardasil®9.

DETAILED DESCRIPTION:
This is a single-center, open-label study on safety, tolerability and immunogenicity of Gardasil®9 in 18 to 45 year-old HIV patients, in 18 to 55 year-old solid-organ transplant (SOT) patients.

This study will enrol 140 HIV patients with CD4+ (cluster of differentiation 4) count of >200cells/mm² and 170 SOT patients, all of whom have not yet received a prophylactic HPV vaccine. The 170 SOT patients will be equally divided over 3 different SOT patient groups, namely heart, lung and kidney transplant patients. Therefore the target is to include approximately 57 heart transplant patients, 57 lung transplant patients and 57 kidney transplant patients. Enrolment in a SOT subgroup will be stopped when 57 patients have been included unless recruitment cannot be achieved within one of the other SOT-patient population.

All enrolled subjects will receive a 3-dose regimen (Day 1, Month 2, and Month 6) of GARDASIL®9. Serum samples will be collected on Day 1 and Month 7 for anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 antibody determination.. The time point for comparison of immune responses will be Month 7, or approximately 4 weeks after the administration of the third dose. The safety/tolerability profile of the vaccine will be evaluated in all subjects in the study. Safety information will be collected on Day 1 through 1 month following the third vaccination or for a total of approximately 7 months for each subject.

The immunogenicity and the safety data will be analyzed per group of patients. More specifically a separate analysis of HIV and SOT patients is planned, since it is expected that the immunosuppressive therapy of SOT patients might have a more profound effect on immunogenicity following vaccination.

This study will provide a comparison of immunogenicity of Gardasil ®9 in immunocompromised patients, with historical controls (15, 18). The number of subjects to be enrolled in the study was determined based on the primary immunogenicity objective.

ELIGIBILITY:
Inclusion Criteria:

1. Independent Ethics Committee (IEC)-approved written informed consent form (ICF) must be obtained from the subject prior to any study-related procedures (including discontinuation of prohibited medication, if applicable) by the subject is given as required by local law.
2. Subject (man or woman) is between the age of 18 years and 0 days and 45 years and 365 days for HIV patients, between 18 years and 0 days and 55 years and 365 days for transplant patients at time of signing the ICF
3. Subject is able to understand and adhere to the study procedures (e.g., is not planning to relocate far from the investigational centre during the study period); is able to read, understand, and complete the vaccination diary; is able to understand the risks involved with the study; and voluntarily agrees to participate in the study by giving written informed consent.
4. * Since the first day of their last menstrual period through Day 1, female subjects have not had sex with males or has had sex with males and used effective contraception with no failures (an example of a failure is a male condom that ruptures during sexual intercourse). Effective contraception is defined as a marketed, approved contraceptive product that the subject has used per the manufacturer's instructions with every act of sexual intercourse. The subject understands and agrees that during the Day 1 through Month 7 period, she should not have sexual intercourse with males without effective contraception. The use of the rhythm method alone, withdrawal alone, and emergency contraception, are not acceptable methods per the protocol. Subjects who have reached menopause, undergone hysterectomy, bilateral oophorectomy, or bilateral tubal ligation are eligible without the use of contraceptives. Postmenopausal status is defined as: (1) No menses for >1 year but <3 years and confirmed by follicle stimulating hormone (FSH) levels elevated into the postmenopausal range, or (2) no menses for at least 3 years.
5. * Subject has had no temperature ≥37.8°C within 24 hours prior to the first injection.
6. Patient considerations

   * HIV patients: have CD4+ T cell count of >200 cells/mm² at the last control (less than 12 months ago).
   * SOT patients received their organ transplantation ≥12 months prior to vaccination and has been stable in the past 6 months (i.e. no acute rejection or other immunological reactions).
7. Apart from having HIV or received a solid organ transplant, the subject is in stable condition (i.e. no graft-versus-host disease or other immunological reactions) and is judged to be in good physical health on the basis of medical history, physical examination (if deemed necessary), and laboratory testing
8. Subject agrees to provide study personnel with a primary telephone number as well as an alternate telephone number for follow-up purposes.

Exclusion Criteria:

1. Subject has a history of an abnormal Pap test or abnormal cervical biopsy results (showing cervical intraepithelial neoplasia or worse) or cervical disease (i.e., surgical treatment for cervical lesions).
2. Subject has history of genital warts, Vulvar Intraepithelial Neoplasia or Vaginal Intraepithelial Neoplasia.
3. Subject has a history of a positive test for HPV.
4. Subject has a history of known prior vaccination with an HPV vaccine, i.e., received a marketed HPV vaccine, or has participated in an HPV vaccine clinical study and has received either active agent or placebo.
5. Subject is pregnant (as determined by serum or urine pregnancy test).
6. Subject is, at the time of signing ICF, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence. Alcohol abusers are defined as those who drink despite recurrent social, interpersonal, and/or legal problems as a result of alcohol use.
7. Subject has a history of severe allergic reaction, including known allergy to any vaccine component, including aluminum, yeast, or BENZONASE® (nuclease, Nycomed [used to remove residual nucleic acids from this and other vaccines]) (e.g., swelling of the mouth and throat, difficulty breathing, hypotension or shock) that met the criteria for serious adverse experiences defined in this protocol.
8. Patient's condition

   1. Exclusion criterion only for HIV patients: Subject has had a splenectomy, or has been diagnosed as having a congenital immunodeficiency, lymphoma, leukaemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune or immunosuppressive condition, or has a history of any disease, which, in the investigator's opinion, may confound the results of the study or pose an additional risk to the subject.
   2. Exclusion criterion only for SOT patients: Subject has had a splenectomy, or has been diagnosed as having a congenital or acquired immunodeficiency, HIV infection, lymphoma, leukaemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory bowel disease, or other autoimmune or immunosuppressive condition, or has a history of any disease, which, in the investigator's opinion, may confound the results of the study or pose an additional risk to the subject.
9. Patient's medication

   1. Exclusion criterion only for HIV patients: Subject is receiving or has received in the year prior to enrolment the following immunosuppressive therapies: radiation therapy, cyclophosphamide, azathioprine, methotrexate, any chemotherapy, cyclosporin, leflunomide (tumour necrosis factor-α antagonists, monoclonal antibody therapies (including rituximab [Rituxan]), intravenous gamma globulin, antilymphocyte sera, or other therapy known to interfere with the immune response. With regard to systemic corticosteroids, a subject will be excluded if she is currently receiving steroid therapy, has recently (defined as within 2 weeks of enrolment) received such therapy, or has received 2 or more courses of high dose corticosteroids (≥20mg/day of prednisone [or equivalent] orally or parenterally) lasting at least 1 week in duration in the year prior to enrolment. Subjects using inhaled, nasal, or topical corticosteroids are considered eligible for the study
   2. Exclusion criterion only for SOT patients: Subject is receiving or has received in the year prior to enrolment the following immunosuppressive therapies: radiation therapy, cyclophosphamide, azathioprine, methotrexate, any chemotherapy, cyclosporin, leflunomide (tumour necrosis factor-α antagonists, monoclonal antibody therapies (including rituximab [Rituxan]) ,intravenous gamma globulin or antilymphocyte sera.
10. Subject has received any immune globulin or blood-derived product within the 3 months prior to the Day 1 vaccination, or plans to receive any such product during Day 1 through Month 7 of the study.
11. Subject has thrombocytopenia or other coagulation disorder that would contraindicate intramuscular injections.
12. * Subject has received inactivated vaccines within 14 days prior to the Day 1 vaccination or has received replicating (live) vaccines within 28 days prior to the Day 1 vaccination. The administration of the inactivated influenza vaccine is allowed 7 days prior to or after each study vaccine.
13. Subject is concurrently enrolled in a clinical study of investigational agent.
14. Subject has a history or current condition of which the investigator believes that it might interfere with the study vaccines.
15. Subject has a history or current evidence of any condition, therapy, lab abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.
16. Subject is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or Sponsor staff directly involved with this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 271 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Vandermeulen, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a single center, open-label, investigator-initiated phase III study (protocol V503-044-IC, NCT03525210) in HIV patients and SOT recipients One hundred HIV patients (age: 18-45 years) and 171 SOT (kidney, heart, lung transplant) patients (age: 18-55 years) were enrolled between April 2018 and January 2019 in the outpatient clinic of the University Hospitals Leuven, Belgium
Period: Overall Study
Arm/Group | HIV Patients | SOT Patients
Started | 100 | 171
Completed | 96 | 169
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Patients | SOT Patients | Total
Number analyzed (Participants) | 100 | 171 | 271
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 171 | 271
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [18 to 45] | 46 [19 to 55] | 42 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 53 | 68
  Male | 85 | 118 | 203
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 2 | 25
  White | 68 | 168 | 236
  More than one race | 9 | 1 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 100 | 171 | 271

OUTCOME MEASURES:

1. Primary Outcome: Seroconversion Following 3 Doses of 9-valent HPV Vaccines
Description: Seroconversion rates of neutralizing antibodies against each HPV vaccine genotypes (6/11/16/18/31/33/45/52/58) one month after completion of a three doses schedule (0, 2 and 6 months) in patients seronegative at baseline for these antibodies.
Time Frame: 7 months (for each subject)
Population: were seronegative to the appropriate HPV type at Day 1, had serology results based on acceptable day ranges and had no protocol deviations that could interfere with the subject's vaccine as judged by the principal investigator.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- HIV Patients: All HIV patients will receive the study vaccines
  9-valent HPV vaccine: Vaccination
  Number and proportion of patients with adverse events.
- SOT Patients: All SOT patients will receive the study vaccines
  9-valent HPV vaccine: Vaccination
  Number and proportion of patients with adverse events.
Arm/Group | HIV Patients | SOT Patients
Number analyzed (Participants) | 91 | 155
Percentage of participants
  Anti-HPV6 | 100 [94.2 to 100] | 64.2 [55.8 to 72.2]
  Anti-HPV11 | 100 [95.3 to 100] | 70.7 [62.7 to 77.8]
  Anti-HPV 16 | 100 [94.3 to 100] | 69.1 [61.0 to 76.4]
  Anti-HPV 18 | 100 [94.6 to 100] | 51.5 [43.2 to 64.0]
  Anti-HPV 31 | 100 [94.4 to 100] | 55.9 [47.6 to 64.0]
  Anti-HPV 33 | 100 [95.1 to 100] | 66.9 [58.8 to 74.3]
  Anti-HPV 45 | 100 [95.3 to 100] | 46.0 [37.8 to 54.3]
  Anti-HPV 52 | 100 [95.8 to 100] | 65.3 [57.1 to 72.9]
  Anti-HPV 58 | 100 [94.9 to 100] | 72.0 [64.1 to 79.0]

2. Secondary Outcome: Adverse Reactions Following 9-valent HPV Vaccination
Description: Number and percentage of subjects with local and systemic sollicited (up to 7 days following each vaccination) and unsollicited adverse events (up to 1 month after the 3rd HPV vaccine) will be analysed
Time Frame: 7 months (for each subject)
Population: Patients with HIV or solid organ transplant who received at least one study vaccine and had at least one follow-up visit for AEs.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Patients | SOT Patients
Number analyzed (Participants) | 99 | 170
Participants | 99 | 170

ADVERSE EVENTS:
Time Frame: Time frame: 7 months
Groups:
- HIV Patients: All HIV patients will receive the study vaccines
  9-valent HPV vaccine: Vaccination
  Number and percentage of patients with adverse events. One patient stopped after the first dose and no safety information could be retrieved.
- SOT Patients: All SOT patients will receive the study vaccines
  9-valent HPV vaccine: Vaccination
  Number and percentage of patients with adverse events. One patient stopped after the first dose and no safety information could be retrieved.
Arm/Group | HIV Patients | SOT Patients
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/170
Serious Adverse Events (participants affected / at risk) | 3/99 | 28/170
Other Adverse Events (participants affected / at risk) | 80/99 | 127/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | HIV Patients (N=99) | SOT Patients (N=170)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Burn-out (Social circumstances) | 1 (1) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Fracture tibia plateau (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abbdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever without focus (Infections and infestations) | 0 (0) | 1 (1)
Gastro-intestinal infections (Infections and infestations) | 0 (0) | 7 (7)
Respiratory infections (Infections and infestations) | 0 (0) | 10 (10)
Skin infections (Infections and infestations) | 0 (0) | 2 (2)
Generalized infections (Infections and infestations) | 0 (0) | 2 (2)
Urogenital infection (Infections and infestations) | 0 (0) | 3 (3)
Acute rejection transplant organ (Immune system disorders) | 0/0 (0) | 1 (1)
dysregulation glycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Relapse renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 1 (1)
Arthrosis neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cyst in transplant kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hemorrhage in adenohypophysis macroadenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pathology of the kidney (Renal and urinary disorders) | 0 (0) | 2 (2)
Respiratory pathology (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Ischemic stroke (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV Patients (N=99) | SOT Patients (N=170)
Injection site pain (General disorders) | 67 (67) | 93 (93)
Injection site swelling (General disorders) | 7 (7) | 14 (14)
injection site erythema (General disorders) | 10 (10) | 10 (10)
Headache (Nervous system disorders) | 9 (9) | 14 (14)

LIMITATIONS AND CAVEATS:
No healthy control group was included in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT03525210/Prot_SAP_000.pdf